CLINICAL TRIAL: NCT04946799
Title: Application of Blood Flow Restriction Training in the Exercise Intervention of Chronic Diseases
Brief Title: The Effect of Blood Flow Restriction Training on Glycemic Control Among Type 2 Diabetes Patients
Acronym: BLFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Nanjing Sport Institute (Unknown); Nanjing Maigaoqiao Community Health Service Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HK-LLWYH-202002
Record Dates: First submitted 2021-05-31; First posted 2021-07-01 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
Keywords: blood flow restriction training; type 2 diabetes; aerobic exercise; randomized-controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-intensity training combined with blood flow restriction group (LI-BFR) (Experimental)
  Interventions: Behavioral: Low-intensity training combined with blood flow restriction (LI-BFR)
- High-intensity aerobic exercise group (HI) (Active Comparator)
  Interventions: Behavioral: High-intensity aerobic exercise (HI)
- Low intensity group (LI) (Placebo Comparator)
  Interventions: Behavioral: Low intensity exercise (LI)

INTERVENTIONS:
Behavioral: Low-intensity training combined with blood flow restriction (LI-BFR) — Participants (n=20) receives low intensity exercise intervention on a cycle ergometer (at 40% of heart rate reserve), with compression belts attached on both thighs, during exercise the belts are inflated with 50% of the participant's arterial occlusion pressure. Exercise is conducted during daytime, 3 times per week, for 12 weeks at Nanjing Maigaoqiao Community Health Service Center. Each exercise session contains 6 sections, each section lasts for 5 minutes, followed with a 1-minute rest period. The compression belt is deflated during the rest period. At least two trained research assistants supervise the exercise in each session. Instant heart rate during exercise is measured with heart rate monitor for each participant.
  Arms: Low-intensity training combined with blood flow restriction group (LI-BFR)
Behavioral: High-intensity aerobic exercise (HI) — Participants (n=20) receives high intensity aerobic exercise intervention on a cycle ergometer (at 70% of heart rate reserve). Exercise is conducted during daytime, 3 times per week, for 12 weeks at Nanjing Maigaoqiao Community Health Service Center. Each exercise session contains 6 sections, each section lasts for 5 minutes, followed with a 1-minute rest period. At least two trained research assistants supervise the exercise in each session. Instant heart rate during exercise is measured with heart rate monitor for each participant.
  Arms: High-intensity aerobic exercise group (HI)
Behavioral: Low intensity exercise (LI) — Participants (n=20) receives low intensity exercise intervention on a cycle ergometer (at 40% of heart rate reserve). Exercise is conducted during daytime, 3 times per week, for 12 weeks at Nanjing Maigaoqiao Community Health Service Center. Each exercise session contains 6 sections, each section lasts for 5 minutes, followed with a 1-minute rest period. At least two trained research assistants supervise the exercise in each session. Instant heart rate during exercise is measured with heart rate monitor for each participant.
  Arms: Low intensity group (LI)

SUMMARY:
Blood flow restriction training (BFRT) combined with resistance or aerobic exercise has been shown to improve the glucose uptake in humans. In addition, BFRT represents a low-load, alternative exercise program for type 2 diabetes patients who often have reduced physical fitness. However, it is not clear to what extent could BFRT improve glycemic control among patients with type 2 diabetes. This pilot randomized-controlled trial aims to investigate the effect of a 12-week, low-intensity BFRT on glycemic control among patients with type 2 diabetes, compared to medium-high intensity aerobic exercise or low-intensity exercise without BFRT.

DETAILED DESCRIPTION:
Objectives:

The pilot randomized study aims to explore the effects of blood flow restriction combined with aerobic training (BFRT) on the glucose and lipid metabolism indexes and vascular endothelial factors of type 2 diabetes, by comparing it with traditional low-intensity and high-intensity aerobic training. It aims to evaluate the effectiveness of BFRT in glycemic control of type 2 diabetes patients.

Study Population:

A total of 60 patients with type 2 diabetes who are 50-65 years old at the Maigaoqiao Community Health Service Center, Qixia District, Nanjing, China, with a course of type 2 diabetes of 2-10 years will be included as the participants.

Randomization:

Participants will be stratified by baseline hemoglobin A1c (HbA1c) and age, they will be randomly assigned into three groups with a block size of six. The study groups are: 1) low-intensity training combined with blood flow restriction group (LI-BFR group, 40% heart rate reserve combined with 50% arterial occlusion pressure, n=20) 2)high-intensity aerobic exercise group (HI group, 70% heart rate reserve, n=20) 3) Low-intensity group (LI group, 40% heart rate reserve, n=20).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes patients diagnosed by at least one of these criteria: 1) random blood glucose >= 11.1mmol/L; 2) fasting blood glucose >= 7.0 mmol/L; 3) 2-hr post oral glucose tolerance test blood glucose >= 11.1mmol/L; 4) hemoglobin A1c >= 6.5%.
* aged between 50-65 years at baseline
* disease course of type 2 diabetes between at least 1 year

Exclusion Criteria:

* type 1 diabetes
* fasting blood glucose > 16.7 mmol/L, or suffers frequent hypoglycemia, or have significant glucose fluctuations considered by the physician
* body mass index > 33 kg/m2
* severe diabetes complications, including cardiovascular diseases, cerebrovascular diseases, diabetic retinopathy, kidney diseases, diabetic ketoacidosis, and diabetic foot ulcers
* neuromuscular disorders, sarcopenia, severe osteoporosis, dementia
* have regular moderate-intensive exercise habit
* resting systolic blood pressure >= 160 mmHg or resting diastolic blood pressure >= 100 mmHg
* abnormal electrocardiogram
* other comorbidities or medications irrelevant to diabetes treatment that may influence glycemia during the past 6 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Fasting glucose at baseline | At baseline, within 7 days before the intervention (observation) starts
  blood glucose level following overnight (12-h) fasting
Fasting glucose at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  blood glucose level following overnight (12-h) fasting
Hemoglobin A1c (HbA1c) at baseline | At baseline, within 7 days before the intervention (observation) starts
  HbA1c level in blood
Hemoglobin A1c (HbA1c) at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  HbA1c level in blood
Fasting insulin at baseline | At baseline, within 7 days before the intervention (observation) starts
  blood insulin level following overnight (12-h) fasting
Fasting insulin at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  blood insulin level following overnight (12-h) fasting

SECONDARY OUTCOMES:
Continuous glucose monitoring | At baseline, within 14 days before the intervention (observation) starts, measurement lasts for 14 days
  14-day continuous glucose monitoring with portable device
Total sleep duration and total awakening duration at baseline | At baseline, within 14 days before the intervention (observation) starts, measurement lasts for at least 7 days
  total sleep duration (in minutes) and total awakening duration after sleep onset (in minutes) assessed by wrist actigraphy (GT3x, Actigraph LLC, Pensacola, FL, USA)
Total sleep duration and total awakening duration at follow-up | At week 13, within 14 days after the completion of the 12-week intervention (observation), measurement lasts for at least 7 days
  total sleep duration (in minutes) and total awakening duration after sleep onset (in minutes) assessed by wrist actigraphy (GT3x, Actigraph LLC, Pensacola, FL, USA)
Pittsburg sleep quality index (PSQI) at baseline | At baseline, within 7 days before the intervention (observation) starts
  Pittsburg sleep quality index global (0-21) and sub-scores (0-3), higher score means poorer quality
Pittsburg sleep quality index (PSQI) at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  Pittsburg sleep quality index global (0-21) and sub-scores (0-3), higher score means poorer quality
Height at baseline | At baseline, within 7 days before the intervention (observation) starts
  height in meters
Height at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  height in meters
Weight at baseline | At baseline, within 7 days before the intervention (observation) starts
  weight in kilograms
Weight at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  weight in kilograms
total cholesterol at baseline | At baseline, within 7 days before the intervention (observation) starts
  total cholesterol level in blood following overnight (12-h) fasting
total cholesterol at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  total cholesterol level in blood following overnight (12-h) fasting
triglyceride at baseline | At baseline, within 7 days before the intervention (observation) starts
  triglyceride level in blood following overnight (12-h) fasting
triglyceride at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  triglyceride level in blood following overnight (12-h) fasting
non-esterified fatty acid (NEFA) at baseline | At baseline, within 7 days before the intervention (observation) starts
  morning NEFA level in blood following overnight (12-h) fasting
non-esterified fatty acid (NEFA) at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  morning NEFA level in blood following overnight (12-h) fasting
IL-6 at baseline | At baseline, within 7 days before the intervention (observation) starts
  morning interleukin-6 level in blood following overnight (12-h) fasting
IL-6 at follow-up | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  morning interleukin-6 level in blood following overnight (12-h) fasting
International Physical Activity Questionnaire - Short Form at baseline | At baseline, within 7 days before the intervention (observation) starts
  International Physical Activity Questionnaire (IPAQ) - Short Form for assessing level of physical activity. Level of physical activity are calculated into metabolic equivalent minutes per week (MET mins/wk) according to the answers of the questionnaire. Higher MET mins/wk refers to higher level of physical activity.
International Physical Activity Questionnaire - Short Form at baseline | At week 13, within 7 days after the completion of the 12-week intervention (observation)
  International Physical Activity Questionnaire (IPAQ) - Short Form for assessing level of physical activity. Level of physical activity are calculated into metabolic equivalent minutes per week (MET mins/wk) according to the answers of the questionnaire. Higher MET mins/wk refers to higher level of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhao, MD, PhD, Principal Investigator — Nanjing Sport Institute; Xiao Tan, PhD, Study Director — Uppsala University
Locations (1):
- Nanjing Maigaoqiao Community Healthcare Center, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No